CLINICAL TRIAL: NCT01052805
Title: Anatomy Study in Control Nerve From Normal Human
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200912006R
Record Dates: First submitted 2010-01-18; First posted 2010-01-20 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2011-10

CONDITIONS: Anatomy of Normal Human Nerves; Microscopic Study; Myelinated Nerve and Unmyelinated Nerve Study
Keywords: nerve; myelinated nerve; unmyelinated nerve

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: nerve from cadaveric donor nerve from nerve graft operation patient
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- harvest nerve: harvest nerve from cadaveric donor and patients receiving nerve graft operation
  Interventions: Procedure: harvest nerve

INTERVENTIONS:
Procedure: harvest nerve — harvest nerve from cadaveric donor and patients receiving nerve graft operation

SUMMARY:
1. To explore the pathology of nerve, vasculature in the normal control nerve
2. Compare the pathology of control nerve and nerve from amputated limb of diabetes

DETAILED DESCRIPTION:
Diabetic foot occurs in 15% of diabetic population (3) and 15% of the diabetic foot patients end up with lower limb amputation. Peripheral neuropathy (sensory, motor and autonomic), peripheral vascular disease, trauma, infection and poor wound healing all contribute to diabetic foot problem.

Peripheral neuropathy could be evaluated in a variety of ways, including vibratory thresholds, thermal thresholds, pressure perception thresholds, muscle strength. All these predict foot ulceration to some degree(1). Motor nerve conduction velocity is an independent predictor for the development of new foot ulcer in diabetic population.

For more detailed structural study of neuropathy in diabetic patient, we could use skin biopsy method. Skin biopsy with PGP9.5 immunohistochemistry has been demonstrated by ultrastructural studies to label the terminal portions of both small myelinated and unmyelinated nerve in the epidermis (5). Intra-epidermal nerve fiber (IENF) density is reduced in patient with impaired glucose tolerance and clinically overt diabetes (5). Previous IENF density study was performed in diabetic patients with sensory symptom but no foot ulcer. Now we tried to evaluate IENF density in severe diabetic foot patient who received below knee amputation. Skin biopsy will be performed at amputated leg. The skin biopsy area will be located at lateral side of distal leg, 10 cm above the lateral malleolus as previous protocol of our group (6). Underlying sural nerve and posterior tibial nerve will be also harvested for further ultra-structural study.

We had previous IRB for "Pathology of skin, nerve and vasculature in the amputated limb of diabetes". However, pathology of normal control nerve is important to compare the pathology of nerve from amputated limb of diabetes. For parotid cancer patients receiving radical parotidectomy, facial nerve is frequently sacrificed. Sural nerve is frequently harvested for reconstruction. Sural nerve is also frequently used in ther nerve construction surgery. During these operations, we could harvested 2 cm more sural nerve for normal nerve pathology study. For cadaveric donor patient, we also could harvest normal nerve for control study.

ELIGIBILITY:
Inclusion Criteria:

* Cadaveric donor
* Patients receiving nerve graft operation

Exclusion Criteria:

* Patient with neurologic disease

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: cadaveric donor patients receiving nerve graft operation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Hsien Hsieh, MD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan